CLINICAL TRIAL: NCT04725162
Title: Epileptogenic Focus Localization for Children With Epilepsy Using 18F-FDG PET Molecular Imaging
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-862
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Peidatrics; Positron emission tomography (PET)
MeSH Terms: conditions — Epilepsy | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epilepsy patients: Pediatric patients with focal epilepsy.
  Interventions: Radiation: 18F-FDG
- Control: Age-matched controls who underwent 18F-FDG PET/CT examination for diseases outside brains.
  Interventions: Radiation: 18F-FDG
- Validation: Children who underwent 18F-FDG PET/MRI to examine extracranial tumors.
  Interventions: Radiation: 18F-FDG

INTERVENTIONS:
Radiation: 18F-FDG — All subjects received 18F-FDG PET examination.

SUMMARY:
This retrospective study aimed to develop a new approach for automatic localization of epilepsy foci in children with epilepsy.

DETAILED DESCRIPTION:
This retrospective study aimed to develop a new approach for automatic localization of epilepsy foci in children with intractable epilepsy.

Pediatric patients with intractable epilepsy would be retrospectively included in this study. The inclusion criteria included (1) age between 6 and 18 y; (2) detailed seizure semiology evaluation, MRI, EEG and interictal 18F-FDG PET/CT examination; (3) clinical diagnosis as focal epilepsy. The exclusion criteria included (a) any history of central nervous system disease; (b) poor image quality due to head movement.

ELIGIBILITY:
Inclusion Criteria:

* 1. age between 6 and 18 years.
* 2. detailed presurgical evaluation, including seizure semiology evaluation, MRI, EEG and interictal 18F-FDG PET/Computer Tomography (CT) examination.
* 3. clinical diagnosis as focal epilepsy.

Exclusion Criteria:

* 1. any history of central nervous system (CNS) disease such as trauma and CNS tumor.
* 2. poor image quality due to head movement.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 130 pediatric patients with focal epilepsy, 67 age-matched controls, and 37 validation group children.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Accuracy | Through study completion, about 6 months
  The accuracy of epilepsy focus localization.
Kappa | Through study completion, about 6 months
  The agreement between experiment result and clinical diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang T, Li Y, Zhao S, Xu Y, Zhang X, Wu S, Dou X, Yu C, Feng J, Ding Y, Zhu J, Chen Z, Zhang H, Tian M. High-resolution pediatric age-specific 18F-FDG PET template: a pilot study in epileptogenic focus localization. Eur J Nucl Med Mol Imaging. 2022 Apr;49(5):1560-1573. doi: 10.1007/s00259-021-05611-w. Epub 2021 Nov 8. PMID 34746970